CLINICAL TRIAL: NCT02913664
Title: Exercise and Intensive Vascular Risk Reduction in Preventing Dementia
Brief Title: Risk Reduction for Alzheimer's Disease
Acronym: rrAD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Health Resources (Other); University of Kansas Medical Center (Other); Washington University School of Medicine (Other); Pennington Biomedical Research Center (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, Rong Zhang, Professor of Neurology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: RZNIA60
Record Dates: First submitted 2016-09-14; First posted 2016-09-26 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Cognitively Normal Older Adults; Hypertension; Subjective Cognitive Decline; Family History of Alzheimer's Disease
Keywords: Dementia; Alzheimer's Disease; Cognitive Function; Blood Pressure; Cholesterol; Physical Activity; Exercise; Magnetic Resonance Imaging
MeSH Terms: conditions — Hypertension; Dementia; Alzheimer Disease; Motor Activity | interventions — Angiotensin Receptor Antagonists; Losartan; Calcium Channel Blockers; Amlodipine; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic Exercise (Ex) (Experimental): Aerobic exercise training; blood and cholesterol management will be standard-care by participant's regular doctor.
  Interventions: Behavioral: Aerobic Exercise Training; Other: Usual Care
- Intensive Reduction of Vascular Risk Factors (IRVR) (Experimental): Lowering SBP < 130 mmHg, administration of atorvastatin 80 mg daily, and stretching exercise.
  Interventions: Drug: Angiotensin II receptor blocker (ARB, losartan) and calcium channel blocker (CCB, amlodipine); Behavioral: Stretching Exercise
- IRVR+Ex (Experimental): A combination of IRVR and aerobic exercise training.
  Interventions: Drug: Angiotensin II receptor blocker (ARB, losartan) and calcium channel blocker (CCB, amlodipine); Behavioral: Aerobic Exercise Training
- Usual Care (Placebo Comparator): Blood and cholesterol management will be standard-care by participant's regular doctor, and stretching exercise.
  Interventions: Other: Usual Care; Behavioral: Stretching Exercise

INTERVENTIONS:
Drug: Angiotensin II receptor blocker (ARB, losartan) and calcium channel blocker (CCB, amlodipine) — Angiotensin II receptor blocker (ARB, losartan) and calcium channel blocker (CCB, amlodipine) will be used to reduce SBP<130 mmHg; atorvastatin 80 mg daily will be administered to reduce blood lipid level. Additional antihypertensives may be used if needed.
  Intensive Reduction of Vascular Risk Factors (IRVR)
  Arms: IRVR+Ex; Intensive Reduction of Vascular Risk Factors (IRVR)
Behavioral: Aerobic Exercise Training — Participants will take part in a supervised, moderate to vigorous aerobic exercise training program for approximately 24 months. This program consists of exercising 3 times per week for about 30 minutes per session at the beginning, and will increase to 4-5 times per week, 40-50 minutes per session over a period of 4-5 months. Exercise frequency, intensity and duration will be maintained at this level during the rest of the study period.
  Arms: Aerobic Exercise (Ex); IRVR+Ex
Other: Usual Care — Participants will follow their regular doctor's recommendations for blood pressure and lipid control.
  Arms: Aerobic Exercise (Ex); Usual Care
Behavioral: Stretching Exercise — Participants will perform home-based stretching exercise 3 times per week, gradually increased to 4-5 times per week over a period of 4-5 months, and maintained at this level during the rest of the study period. They will be encouraged to attend monthly stretching exercise classes, which will be led by study staff or exercise trainers.
  Arms: Intensive Reduction of Vascular Risk Factors (IRVR); Usual Care

SUMMARY:
Physical inactivity, high blood pressure and dyslipidemia are risk factors for Alzheimer's disease (AD) and vascular dementia. Importantly, these risk factors are modifiable with lifestyle changes, pharmacological treatment, or both. The rrAD study will determine effects of aerobic exercise training and intensive vascular risk reduction on cognitive performance in older adults who have high risk for AD.

DETAILED DESCRIPTION:
Numerous lines of evidence suggest that interventions that confer therapeutic benefits for cardiovascular health are also associated with improvements in, or preservation of, cognitive function. Many believe "What's good for the heart is good for the brain." However, stronge scientific evidence is needed to prove this hypothesis. The rrAD study is a 4-arm, multicenter, randomized trial to assess the effects of aerobic exercise training and intensive pharmacological reduction of vascular risk factors on cognitive performance in older adults who have high risk for AD, that is, those who have high blood pressure, family history of dementia or subjective memory complaints. Furthermore, rrAD will examine effects of exercise and vascular risk reduction on brain volume, perfusion, and neural network connectivity using magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Age 60-85, all races/ethnicities, and both sexes are eligible.
2. a) A positive family history of dementia defined as having at least one first-degree relative with a history of AD or other type of dementia,or b) having subjective cognitive decline.
3. Mini-Mental State Exam (MMSE) ≥ 26 to exclude gross dementia.
4. Must lead a sedentary lifestyle defined by not having an "active" rating on Rapid Assessment of Physical Activity (RAPA), i.e., score below 6 on RAPA.
5. a) Individuals treated for HTN with 110 ≤ SBP ≤ 130 mmHg; or b) Individuals with SBP > 130 and SBP < 180 (If an individual, not treated for HTN, has a SBP ≥ 125 mmHg, consider rescreening after 24 hours).
6. Willingness to be randomized into the treatment groups and ability to return to clinic for follow-up visits over 24 months.
7. Fluency in English, adequate visual and auditory acuity to allow neuropsychological testing.
8. Participants must have a regular healthcare provider.
9. Physical ability to undergo exercise training; able to walk 10 minutes without pain.

Exclusion Criteria:

1. Clinically documented history of stroke, focal neurological signs or other major cerebrovascular diseases based on clinical judgment or MRI/CT scans such as evidence of infection, infarction or other brain lesions.
2. Diagnosis of AD or other type of dementia, or significant neurologic diseases such as Parkinson's disease, seizure disorder, multiple sclerosis, history of severe head trauma or normal pressure hydrocephalus.
3. Evidence of severe major depression (GDS > 12, may be rescreened after 12 weeks or longer if evidence of reactive depression or temporary mood disturbances) or clinically significant psychopathology(e.g. psychosis and schizophrenia); if hospitalized in past year, can be rescreened in 6 months; or presence of a major psychiatric disorder that in the investigator's opinion, could interfere with adherence to research assessments or procedures.
4. Unstable heart disease based on clinical judgment (e.g., heart attack/cardiac arrest, cardiac bypass procedures within previous 6 months and congestive heart failure),or other severe medical conditions.
5. History of atrial fibrillation and evidence on ECG with any of the following: active symptoms of persistent palpitation, dizziness, history of syncope, chest pain, dyspnea, orthopnea, shortness of breath at rest, or paroxysmal nocturnal dyspnea within the past 6 months; resting heart rate of < 30 or > 110 bpm; taking class I or III anti-arrhythmic drugs including flecanide, propafenone, dronedarone, sotalol, dofetilide, and amiodarone; or clinical concerns for safely participating in exercise and lowering blood pressure.
6. Systolic BP equal or greater than 180 mmHg and/or diastolic BP equal or greater than 110 mmHg, may be rescreened in 1 week.
7. Orthostatic hypotension, defined as the third standing SBP < 100mmHg, may be rescreened after 2 weeks.
8. History of significant autoimmune disorders such as systemic lupus erythematosus, rheumatoid arthritis, or polymyalgia rheumatic.
9. Significant history of alcoholism or drug abuse within the last five years.
10. Uncontrolled diabetes mellitus, defined as hemoglobin A1C > 7.5%, or requiring insulin treatment.
11. Regularly smoking cigarette within the past year.
12. Women with a potential for pregnancy, lactation/child bearing (2 year post- menopausal or surgically sterile to be considered not child bearing potential).
13. Participant enrolled in another investigational drug or device study, either currently or within the past 2 months.
14. Severe obesity with BMI ≥ 45; clinical judgment should be applied in all cases to assess patient safety and anticipated compliance.
15. Allergy to angiotensin receptor blockers (ARBs), i.e., drugs that have a suffix "-sartan".
16. Allergy to other study drugs or their ingredients; for example, clinical history or self-reported allergy or intolerance to atorvastatin.
17. Abnormal screening laboratory tests (e.g., liver ALT and AST > 3 x ULN, CK > 3 x ULN, GFR < 30 or Hct < 28%); may be rescreened after 2 weeks or longer.
18. A medical condition likely to limit survival to less than 3 years.
19. Participant has any condition(s) judged by the study investigator to be medically inappropriate, risky or likely to cause poor study compliance. For example:

    1. Plans to move outside the clinic catchment area in the next 2 years;
    2. Significant concerns about participation in the study from spouse, significant other, or family members;
    3. Lack of support from primary health care provider;
    4. Residence too far from the study clinic site such that transportation is a barrier including persons who require transportation assistance provided by the study clinic funds for screening or randomization visits;
    5. Residence in a nursing home; persons residing in an assisted living or retirement community are eligible if they meet the other criteria.
    6. Other medical, psychiatric, or behavioral factors that, in the judgment of the site PI or clinician, may interfere with study participation or the ability to follow the study Protocol.
    7. Couples or significant partners who live together cannot be enrolled or participate simultaneously in the study.
20. Lack of approval from participant's regular healthcare providers, i.e. a signed letter of agreement for the participants to be enrolled in rrAD.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in global neurocognitive function | 2 Years
  Alzheimer's Disease Cooperative Study-Preclinical Alzheimer Cognitive Composite (ADCS-PACC) and NIH Toolbox (NIH-TB) Cognition Battery will be used to assess changes in neurocognitive function. The composite z-score for global cognition will be obtained by conversion of individual test scores to the standardized z-scores, then averaged to obtain a composite score.

SECONDARY OUTCOMES:
Domain-specific neurocognitive function assessed by using the tests included in the ADCS-PACC and NIH-TB Cognition. | 2 Years
Whole brain and hippocampal volume assessed via Magnetic Resonance Imaging (MRI). | 2 years
Global and regional brain perfusion assessed via Magnetic Resonance Imaging (MRI). | 2 years
Brain white matter hyperintensity (WMH) assessed via Magnetic Resonance Imaging (MRI). | 2 years
Brain white matter microstructural integrity assessed via Magnetic Resonance Imaging (MRI). | 2 years
Brain neural network functional connectivity assessed via functional Magnetic Resonance Imaging (MRI). | 2 years
Patient-reported outcomes (PRO) of mental and physical health and health-related quality of life assessed by using NIH PROMIS. | 2 years
Physical function assessed via the Short Physical Performance Battery (SPPB). | 2 years
Dual task performance assessed via distracted and non-distracted 10 meter walk. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rong Zhang, PhD, Principal Investigator — University of Texas Southwestern Medical Center; Jeffrey Keller, PhD, Principal Investigator — Pennington Biomedical Research Center; Jeffrey Burns, MD, Principal Investigator — University of Kansas Medical Center; Ellen Binder, MD, Principal Investigator — Washington University School of Medicine; Munro Cullum, PhD, Principal Investigator — UT Southwestern; Diana Kerwin, MD, Principal Investigator — Texas Health Resources
Locations (4):
- United States (4):
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Washington University in St. Louis, St Louis, Missouri
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will be shared approximately 18-24 months after the primary study publication.

REFERENCES:
- [Derived] Szabo-Reed A, Clutton J, White S, Van Sciver A, White D, Morris J, Martin L, Lepping R, Shaw A, Puchalt JP, Montgomery R, Mahnken J, Washburn R, Burns J, Vidoni ED. COMbined Exercise Trial (COMET) to improve cognition in older adults: Rationale and methods. Contemp Clin Trials. 2022 Jul;118:106805. doi: 10.1016/j.cct.2022.106805. Epub 2022 May 27. PMID 35636733
- [Derived] Vidoni ED, Kamat A, Gahan WP, Ourso V, Woodard K, Kerwin DR, Binder EF, Burns JM, Cullum M, Hynan LS, Vongpatanasin W, Zhu DC, Zhang R, Keller JN. Baseline Prevalence of Polypharmacy in Older Hypertensive Study Subjects with Elevated Dementia Risk: Findings from the Risk Reduction for Alzheimer's Disease Study (rrAD). J Alzheimers Dis. 2020;77(1):175-182. doi: 10.3233/JAD-200122. PMID 32716358
- [Derived] Gottesman RF. To INFINITY and Beyond: What Have We Learned and What Is Still Unknown About Blood Pressure Lowering and Cognition? Circulation. 2019 Nov 12;140(20):1636-1638. doi: 10.1161/CIRCULATIONAHA.119.042827. Epub 2019 Nov 11. No abstract available. PMID 31710528
- [Derived] Szabo-Reed AN, Vidoni E, Binder EF, Burns J, Cullum CM, Gahan WP, Gupta A, Hynan LS, Kerwin DR, Rossetti H, Stowe AM, Vongpatanasin W, Zhu DC, Zhang R, Keller JN. Rationale and methods for a multicenter clinical trial assessing exercise and intensive vascular risk reduction in preventing dementia (rrAD Study). Contemp Clin Trials. 2019 Apr;79:44-54. doi: 10.1016/j.cct.2019.02.007. Epub 2019 Mar 1. PMID 30826452
- See also: Study Website — http://www.rradtrial.org/